CLINICAL TRIAL: NCT00344773
Title: An Open-label, Multi-centre Study to Evaluate Efficacy and Safety of Gefitinib as the First-line Treatment for Locally Advanced (IIIB), Metastatic (IV) or Recurrent Pulmonary Adenocarcinoma Patients With Epidermal Growth Factor Receptor (EGFR) Mutation.
Brief Title: First-line Treatment for Adenocarcinoma Patients With Epidermal Growth Factor Receptor (EGFR) Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7913L00056
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Results first posted 2010-06-04 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Pulmonary Cancer
Keywords: Locally advanced (IIIB) pulmonary adenocarcinoma with EGFR mutation; Metastatic (IV) pulmonary adenocarcinoma with EGFR mutation; Recurrent pulmonary adenocarcinoma with EGFR mutation
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis | interventions — Gefitinib

ARMS (1):
- Gefitinib (Experimental): Gefitinib 250mg tablet once daily
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — 250mg tablet oral tablet once daily
  Other Names: ZD1839; IRESSA

SUMMARY:
The purpose of this study is to evaluate the overall objective tumor response rate (ORR) of Gefitinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients require histological biopsy and paraffin block more than 5mg from the original tumour or metastatic site to perform EGFR mutational analysis
* WHO Performance Status 0-2
* No prior chemotherapy, biological or immunological therapy/surgery

Exclusion Criteria:

* Any evidence of clinically active interstitial lung disease
* Newly diagnosed CNS metastases that have not yet been definitively treated with surgery /radiation
* Patients with previously diagnosed and treated CNS metastases or spinal cord compression

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: HyeJong Yoo, Study Director — AstraZeneca
Locations (2):
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul

REFERENCES:
- [Derived] Kim DW, Lee SH, Lee JS, Lee MA, Kang JH, Kim SY, Shin SW, Kim HK, Heo DS. A multicenter phase II study to evaluate the efficacy and safety of gefitinib as first-line treatment for Korean patients with advanced pulmonary adenocarcinoma harboring EGFR mutations. Lung Cancer. 2011 Jan;71(1):65-9. doi: 10.1016/j.lungcan.2010.04.005. PMID 20430469

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 147 patients were screened for epidermal growth factor receptor (EGFR) mutation and 46 patients were enrolled in this study. Subjects were recruited by 7 investigational centers throughout South Korea from Mar 2006 to May 2007
Groups:
- Gefitinib: Gefitinib 250mg tablet
Period: Overall Study
Arm/Group | Gefitinib
Started | 46
Completed | 25
Not Completed | 21
Not completed — Adverse Event | 2
Not completed — Objective Disease Progression | 16
Not completed — Withdrawal by Subject | 1
Not completed — Not Eligible for the study | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gefitinib
Number analyzed (Participants) | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 60 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had an Objective Response Rate(ORR) Based on Response Evaluation Criteria In Solid Tumors (RECIST) Criteria.
Description: Objective Response Rate (ORR) is defined as participants who had complete response (CR) or partial response(PR) divided by the total number of patients.
  RECIST criteria:
  CR = disappearance of all target lesions PR = 30% decrease in the sum of the longest diameter of target lesions PD = 20% increase in the sum of the longest diameter of target lesions SD (stable disease) = small changes that do not meet above criteria
Time Frame: baseline to 12 months
Measure: Number; unit: Percent of Participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 46
Percent of Participants | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival calculated using Kaplan-Meier Product Limit. Median PFS was not able to be calculated because the rate of PFS was below 50% at the end of follow-up period. Therefore, PFS percentage at 4 months is provided.
Time Frame: baseline to 4 months
Measure: Number; unit: Percent of Participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 46
Percent of Participants | 86.25 [0.7191 to 0.9358]

3. Secondary Outcome: Overall Survival (OS)
Description: Median Overal survival was not able to be calculated because the rate of OS was below 50% at the end of follow-up period. Therefore, OS percentage at 12 months is provided.
Time Frame: baseline to 12 months
Measure: Number; unit: Percent of Participants
Arm/Group | Gefitinib
Number analyzed (Participants) | 46
Percent of Participants | 82.26 (0)

4. Secondary Outcome: Safety Profile: Participants With Adverse Events
Description: Safety profile as defined by adverse events and serious adverse events throughtout the study period. Details listed in the SAE and Other AE section.
Time Frame: baseline to end of study
Reporting Status: Not Posted
Measure: Number; unit: participants with adverse events

ADVERSE EVENTS:
Arm/Group | Gefitinib
Serious Adverse Events (participants affected / at risk) | 4
Other Adverse Events (participants affected / at risk) | 44
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Gefitinib
Pneumonia (Infections and infestations) | 2/46
Multiple contusion with Lt.9.10.11th rib fracture (Injury, poisoning and procedural complications) | 1/46
Intramuscular myxoma in the left intraspinatos muscle (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/46
Diarrhea (Gastrointestinal disorders) | 1/46
Myoclonus (Nervous system disorders) | 1/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Gefitinib
Alopecia (Skin and subcutaneous tissue disorders) | 5/46
Anorexia (Metabolism and nutrition disorders) | 17/46
Back-pain (Musculoskeletal and connective tissue disorders) | 4/46
Common cold (Infections and infestations) | 3/46
Constipation (Gastrointestinal disorders) | 7/46
Cough (Respiratory, thoracic and mediastinal disorders) | 13/46
Desquamation (Skin and subcutaneous tissue disorders) | 9/46
Diarrhea (Gastrointestinal disorders) | 16/46
Dizziness (Nervous system disorders) | 5/46
Dry-skin (Skin and subcutaneous tissue disorders) | 3/46
Dyspepsia (Gastrointestinal disorders) | 4/46
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6/46
Epigastric pain (Gastrointestinal disorders) | 3/46
Epigastric soreness (Gastrointestinal disorders) | 3/46
General-weakness (Gastrointestinal disorders) | 3/46
Hand foot syndrome (Skin and subcutaneous tissue disorders) | 3/46
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 3/46
Headache (Nervous system disorders) | 6/46
Indigestion (Gastrointestinal disorders) | 3/46
Itching (Skin and subcutaneous tissue disorders) | 16/46
Mucositis (Skin and subcutaneous tissue disorders) | 3/46
Nausea (Gastrointestinal disorders) | 12/46
Neuropathy (Nervous system disorders) | 4/46
Rash (Skin and subcutaneous tissue disorders) | 3/46
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3/46
Skin-rash (Skin and subcutaneous tissue disorders) | 14/46
Sorethroat (Respiratory, thoracic and mediastinal disorders) | 3/46
Sputum (Respiratory, thoracic and mediastinal disorders) | 10/46
Stomatitis (Gastrointestinal disorders) | 9/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less